CLINICAL TRIAL: NCT01965223
Title: Stereotactic Ablative Fractionated Radiotherapy Versus Radiosurgery for Oligometastatic Neoplasia to the Lung: A Randomised Phase II Trial
Brief Title: A Randomized Phase II Study of Stereotactic Ablative Body Radiotherapy for Metastases to the Lung (TROG 13.01 SAFRON II)
Acronym: SAFRON II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Collaborators: Australasian Lung Cancer Trials Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TROG 13.01; TROG 13.01 (Other: Trans Tasman Radiation Oncology Group); 13001 (Other: Australasian Lung Trials Group); 1111-1136-6607 (Registry Identifier: WHO)
Record Dates: First submitted 2013-10-13; First posted 2013-10-18 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Cancer; Metastases to the Lung
Keywords: Oligometastatic; Neoplasia; Radiosurgery; Stereotactic Ablative Body Radiotherapy; SABR; Metastases to the Lung; Non Haematological
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multi-fraction SABR (Experimental): Radiotherapy: 48Gy delivered in 4 fractions, delivered over 2 weeks, with each fraction delivered 48 hours apart.
  Interventions: Radiation: Multi-fraction SABR
- Single fraction SABR (Experimental): Radiotherapy: 28Gy delivered in 1 fraction
  Interventions: Radiation: Single Fraction SABR

INTERVENTIONS:
Radiation: Multi-fraction SABR — Multi-fraction SABR; 48Gy delivered in 4 fractions, delivered over 2 weeks, with each fraction delivered 48 hours apart.
  Arms: Multi-fraction SABR
Radiation: Single Fraction SABR — Single fraction SABR; 28Gy delivered in 1 fraction
  Arms: Single fraction SABR

SUMMARY:
The main purpose of this study is to determine the safety (defined as number of participants experiencing ≥ 5% toxicity at 12 months post treatment) of stereotactic ablative fractionated radiotherapy versus radiosurgery for oligometastatic neoplasia to the lung.

DETAILED DESCRIPTION:
Stereotactic Ablative Body Radiotherapy (SABR) is an exciting novel radiotherapy technique that is delivered over very few sessions. In the case of limited pulmonary 'oligometastases', SABR can result in long-term survival. It is non-invasive and associated with high rates of tumour control and relatively low toxicity. Additionally, the large doses of precision radiotherapy involved may evoke a strong immune response to recognise and attack any remaining tumour cells. In the future, SABR may be an attractive alternative to invasive surgery. There are two SABR techniques emerging in Australia; fractionated and single fraction treatments. We aim to conduct the first clinical trial of SABR in patients with limited pulmonary metastases testing fractionated versus single fraction treatments.

The primary aim of this study is to evaluate the toxicity, Quality of Life, clinical efficacy and cost effectiveness of single fraction SABR compared to multi-fraction SABR in patients with oligometastases to the lung.

The secondary aim of this study is to assess the immune response evoked by both fractionated and single fraction SABR and its prognostic implications for patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. A maximum of three metastases to the lung from any non-haematological malignancy
2. Tumour diameter ≤5cm
3. Targets are located away from central structures (defined as 2cm beyond bifurcation of lobar bronchi and central airways). Targets in proximity to chest wall and mediastinum that meet these inclusion criteria are eligible.
4. Patients must be medically inoperable, technically high risk or have declined surgery.

Exclusion Criteria:

1. Previous high-dose thoracic radiotherapy.
2. Cytotoxic chemotherapy within 3 weeks of commencement of treatment, or concurrently with treatment. Hormonal manipulation agents are not excluded (e.g. aromatase inhibitors, selective oestrogen receptor modulators, and gonadotrophin releasing hormone receptor modulators)
3. Targeted agents (such as sunitinib and tarceva) within 7 days of commencement of treatment, or concurrently with treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-02-04 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2020-07-27 (Actual)

PRIMARY OUTCOMES:
Toxicity | 12 months
  The primary outcome is safety, defined as number of participants experiencing less than or equal to 5% toxicity at 12 months post treatment (toxicity as measured by CTCAE V4).

SECONDARY OUTCOMES:
Quality of Life | 24 months
  To compare quality of life outcomes between techniques assessed using EQ-5DL and MDASI-LC questionnaires.
Time to local failure | 24 months
  Local progression free survival assesed by CT scan and clinical assessment
Overall survival | 24 months
  Overall survival assesed by clinical assessment
Time to distant failure | 24 months
  Time to distant failure assessed by CT scan and clinical assessment
Resources use and costs associated with treatment | 24 months
  Resources use and costs associated with treatment assessed by EQ5DL and accessing Medicare data
Disease Free Survival | 24 months
  Disease free survival will be measured from the date of randomisation to the date of a local recurrence, regional or distant metastasis, or death from any cause, whichever occurs first.

OTHER OUTCOMES:
Immune response | 3 months
  To explore immune system responses to single fraction and multi-fraction SABR.

CONTACTS AND LOCATIONS:
Overall Officials: Shankar Siva, Study Chair — Peter MacCallum Cancer Centre, Australia
Locations (9):
- Australia (9):
  - Liverpool Hospital, Liverpool, New South Wales
  - Calvary Mater Hospital, Newcastle, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Northern Sydney Cancer Centre (RNS), St Leonards, New South Wales
  - Cambelltown Hospital, Sydney, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Center, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia

REFERENCES:
- [Derived] Siva S, Sakyanun P, Mai T, Wong W, Lim A, Ludbrook J, Bettington C, Rezo A, Pryor D, Hardcastle N, Kron T, Higgs B, Le H, Skala M, Gill S, Eade T, Awad R, Sasso G, Vinod S, Montgomery R, Ball D, Bressel M. Long-Term Outcomes of TROG 13.01 SAFRON II Randomized Trial of Single- Versus Multifraction Stereotactic Ablative Body Radiotherapy for Pulmonary Oligometastases. J Clin Oncol. 2023 Jul 1;41(19):3493-3498. doi: 10.1200/JCO.23.00150. Epub 2023 May 14. PMID 37179526
- [Derived] Siva S, Bressel M, Mai T, Le H, Vinod S, de Silva H, Macdonald S, Skala M, Hardcastle N, Rezo A, Pryor D, Gill S, Higgs B, Wagenfuehr K, Montgomery R, Awad R, Chesson B, Eade T, Wong W, Sasso G, De Abreu Lourenco R, Kron T, Ball D, Neeson P; Stereotactic Ablative Fractionated Radiotherapy Versus Radiosurgery for Oligometastatic Neoplasia to the Lung (SAFRON) II Study Investigators. Single-Fraction vs Multifraction Stereotactic Ablative Body Radiotherapy for Pulmonary Oligometastases (SAFRON II): The Trans Tasman Radiation Oncology Group 13.01 Phase 2 Randomized Clinical Trial. JAMA Oncol. 2021 Oct 1;7(10):1476-1485. doi: 10.1001/jamaoncol.2021.2939. PMID 34455431